CLINICAL TRIAL: NCT07380633
Title: Toripalimab Plus Bevacizumab Combined Three Intra-arterial Therapies (Transarterial Chemoembolization, Hepatic Artery Infusion Chemotherapy, or Transarterial Chemoembolization Plus Hepatic Artery Infusion Chemotherapy) for Unresectable Hepatocellular Carcinoma: a Phase 2, Multicenter Randomised Non-comparative Trial
Brief Title: Toripalimab Plus Bevacizumab Combined Three Intra-arterial Therapies (TACE, HAIC, or TACE-HAIC) for Unresectable Hepatocellular Carcinoma: a Phase 2, Multicenter Randomised Non-comparative Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2025-900-01
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: The TACE was performed using 30 mg/m2 of epirubicin, 300mg/m2 carb mixed with 2-5 mL lipiodol, followed by pure lipiodol. The HAIC regimen at the following dosage: 85 mg/m2 of oxaliplatin infusion for 2 hours; leucovorin, 400 mg/m2 infusion for 2 hours; 400 mg/m2 of 5-FU bolus; and 1200mg/m2 of continuous 5-FU infusion for 23 hours, respectively. TACE-HAIC was performed TACE following by HAIC. Repeated transarterial therapy was performed at intervals of 3-4 weeks. Toripalimab was adminstated at 240mg and bevacizumab was adminstated at 15mg/kg on next day after transarterial therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TACE-HAIC+T-B (Experimental): Transartery chemoembolization and hepatic artery infusion of FOLFOX, simultaneously followed by toripalimab of 240mg plus bevacizumab (15mg/kg)
  Interventions: Drug: TACE-HAIC+T-B
- TACE+T-B (Active Comparator): Transartery chemoembolization followed by toripalimab of 240mg plus bevacizumab (15mg/kg)
  Interventions: Drug: TACE+T-B
- HAIC+T-B (Active Comparator): hepatic artery infusion of FOLFOX regimen followed by toripalimab of 240mg plus bevacizumab (15mg/kg)
  Interventions: Drug: HAIC+T-B

INTERVENTIONS:
Drug: TACE-HAIC+T-B — Transartery chemoembolization and hepatic artery infusion of FOLFOX, simultaneously followed by toripalimab of 240mg plus bevacizumab (15mg/kg)
  Arms: TACE-HAIC+T-B
Drug: HAIC+T-B — FOLFOX-based HAIC regimen followed by toripalimab of 240mg plus bevacizumab
  Arms: HAIC+T-B
Drug: TACE+T-B — TACE was performed using 30 mg/m2 of epirubicin, 300mg/m2 carb mixed with 2-5 mL lipiodol, followed by pure lipiodol, followed by toripalimab was adminstated at 240mg and bevacizumab was adminstated at 15mg/kg.
  Arms: TACE+T-B

SUMMARY:
Toripalimab and bevacizumab (T-B) was approve for unresectable hepatocellular carcinoma (uHCC). Transartial therapies, including transarterial chemoembolization (TACE), hepatic artery infusion chemotherapy (HAIC), and TACE-HAIC are commonly used for uHCC. Increasing evidence showed that combined systemic therapy and transarterial therapy will improve the response rate for those patients. It is unknown whether which tranarterial therapy will proved favorable efficiency when combined T-B. This phase 2 clinical trial aims to investigate the short outcome of T-B with three distinct transarterial therapies for uHCC.

DETAILED DESCRIPTION:
Toripalimab in combination with bevacizumab (T-B) has been approved for the treatment of unresectable hepatocellular carcinoma (uHCC). Transarterial therapies-including transarterial chemoembolization (TACE), hepatic arterial infusion chemotherapy (HAIC), and combined TACE-HAIC-are widely used in the management of uHCC. Growing evidence suggests that combining systemic therapy with transarterial approaches can enhance response rates in these patients. However, it remains unclear which transarterial modality, when used alongside T-B, offers the most favorable efficacy. This phase 2 clinical trial is designed to evaluate and compare the short-term outcomes of T-B in combination with three different transarterial therapies for uHCC.

ELIGIBILITY:
Inclusion Criteria:

* (a) patients were diagnozied with unresectable HCC, (b) Child-Pugh A or B liver function; (d) Eastern Cooperative Oncology Group (ECOG) performance status 0-1; (e) adequate hematologic blood counts (white blood cell count >3ⅹ109/L, absolute neutrophil count >1.5ⅹ109/L, platelet count >10ⅹ109/L, hemoglobin concentration >85 g/L);

Exclusion Criteria:

* (a) severe underlying cardiac, pulmonary, or renal diseases; (b) history of a second primary malignant tumor; (c) contraindication to either toripalimab and bevacizumab.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-23 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
12-Month PFS Rate (Intention-to-Treat) | 12 months
  This measure reports the proportion of all randomized patients (ITT population) who are progression-free at 12 months post-randomization.

SECONDARY OUTCOMES:
OS | 12 months
  overall survival time after randomisation, taking into account all deaths
PFS | 12 months
  progression free survival time after randomisation, taking into account all deaths
ORR | 12 months
  objective response rate assessed by RECIST 1.1
adverse event | 12 months
  adverse event was assessed by NCI-CTC 5.0 to evaluate safety

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No